CLINICAL TRIAL: NCT00096070
Title: Phase II Study of Oxaliplatin, Continuous 5-Fluorouracil and External Beam Radiation Followed by Gemcitabine in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Radiotherapy Combined With Oxaliplatin and Fluorouracil Followed By Gemcitabine in Treating Patients With Locally Advanced, Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01816; N0349; CDR0000391191; NCCTG-N0349; U10CA025224 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Pancreas; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy; Radiation; Oxaliplatin; Fluorouracil; Gemcitabine

ARMS (1):
- Arm I (Experimental): Patients undergo radiotherapy once daily, 5 days a week, for 5.5 weeks. Beginning concurrently with radiotherapy, patients receive oxaliplatin IV over 2 hours on days 1, 15, and 29 and fluorouracil IV continuously for 5.5 weeks. Beginning 4-6 weeks after the completion of chemoradiotherapy, patients receive gemcitabine IV over 30 minutes on days 1 and 8. Treatment with gemcitabine repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: radiation therapy; Drug: oxaliplatin; Drug: fluorouracil; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar

SUMMARY:
This phase II trial is studying how well giving radiation therapy together with oxaliplatin and fluorouracil followed by gemcitabine works in treating patients with locally advanced, unresectable pancreatic cancer. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy, such as oxaliplatin, fluorouracil, and gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Oxaliplatin may also make the tumor cells more sensitive to radiation therapy. Giving radiation therapy with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the 1-year survival rate in patients with locally advanced, unresectable adenocarcinoma of the pancreas treated with concurrent external beam radiotherapy, oxaliplatin, and fluorouracil followed by gemcitabine.

SECONDARY OBJECTIVES:

I. Determine overall survival, time to disease progression, and confirmed response rate in patients treated with this regimen.

II. Determine toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients undergo radiotherapy once daily, 5 days a week, for 5.5 weeks. Beginning concurrently with radiotherapy, patients receive oxaliplatin IV over 2 hours on days 1, 15, and 29 and fluorouracil IV continuously for 5.5 weeks. Beginning 4-6 weeks after the completion of chemoradiotherapy, patients receive gemcitabine IV over 30 minutes on days 1 and 8. Treatment with gemcitabine repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Unresectable disease, including subtotal resection and gross residual disease
  * Locally advanced disease
* No cystadenocarcinoma of the pancreas
* No pancreatic tumors of neuroendocrine origin
* No microscopic residual disease as only evidence of pancreatic cancer
* All disease must be encompassable within standard radiotherapy fields for pancreatic cancer
* No distant metastases (liver or lung metastases or peritoneal spread)

  * No evidence of metastatic disease outside the planned radiotherapy field
* Performance status - ECOG 0-1
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to maintain adequate oral nutrition
* No significant infection
* No significant nausea or vomiting
* No other medical condition that would preclude study participation
* No other malignancy within the past 3 years except nonmelanoma skin cancer, carcinoma in situ of the cervix, or organ-confined prostate cancer (Gleason score < 7)
* No known allergy to platinum compounds
* No prior biologic therapy
* No concurrent biologic therapy
* No concurrent immunotherapy
* No prior chemotherapy
* No other concurrent chemotherapy
* No prior radiotherapy that would overlap planned radiotherapy fields
* No other concurrent radiotherapy
* See Disease Characteristics
* At least 21 days since prior laparotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-12; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
1-year survival rate | At 1 year
  1-year survival will be considered "success". The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. If more than 1 patients is lost to follow-up, we will use Kaplan-Meier estimates for the 6-month and 12-month overall survival rates. 95% confidence intervals for the true success proportion will be calculated according the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Survival time | Time from registration to death due to any cause, assessed up to 3 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Confirmed tumor response, defined to be a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart | Up to 6 months
Time to disease progression | Time from registration to documentation of disease progression, assessed up to 3 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Duration of response | Date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented, assessed up to 3 years
Time to treatment failure | Time from the date of randomization to the date at which the patient is removed from treatment due to progression, toxicity, or refusal, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: George Kim, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States